CLINICAL TRIAL: NCT03965936
Title: Effect of Adipose Derived Stem Cells on Survival of Fat as Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Aliaa Ismail Ali Ismail, principle investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: alexderma 2
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Skin Rejuvenation; Lipofilling
Keywords: adipose tissue derived stem cells; lipofilling

STUDY DESIGN:
Intervention Model Description: split face
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lipofilling (Placebo Comparator): subcutaneous injection of lipoaspiate (microfat) in one temporal region
  Interventions: Procedure: lipofilling
- lipofilling enriched with adipose tissue derived stem cells (Active Comparator): subcutaneous injection of lipoaspiate enriched with adipose tissue derived stem cells in one temporal region
  Interventions: Procedure: lipofilling enriched with adipose tissue derived stem cells

INTERVENTIONS:
Procedure: lipofilling — Under local anesthesia using strict aseptic technique, a small incision will be done in the lateral aspect of the thigh or lower abdomen, through which the infiltration cannula will be introduced to inject the local anesthetic solution using the wet technique. This will be followed 15 minutes later by lipo-aspiration of 75 ml fat ) using a blunt tipped cannula under the negative suction pressure of a 60 ml syringe. 50 ml is used for preparation of microfat. then with blunt cannula,subcutaneous injection of the required volume of microfat is placed into temporal region.
  Arms: lipofilling
Procedure: lipofilling enriched with adipose tissue derived stem cells — Under local anesthesia using strict aseptic technique, a small incision will be done in the lateral aspect of the thigh or lower abdomen, through which the infiltration cannula will be introduced to inject the local anesthetic solution using the wet technique. This will be followed 15 minutes later by lipo-aspiration of 75 ml fat using a blunt tipped cannula under the negative suction pressure of a 60 ml syringe. 50 ml is used for preparation of microfat. 25 ml is used for preparation of autologous adipose tissue derived stem cells (At-ADSCs) using enzymatic digestion and differential centrifugation in the Center of Excellence for Research in Regenerative Medicine and its Application (CERRMA), Alexandria Faculty of Medicine.
  Subcutaneous injection of the required volume of microfat combined with stromal vascular fraction containing adipose tissue derived stem cells, is placed into temporal region.
  Arms: lipofilling enriched with adipose tissue derived stem cells

SUMMARY:
this research is to study the effect of Adipose Derived Stem Cells on Survival of Fat as Filler

DETAILED DESCRIPTION:
Skin aging is a complex biological process.The physiological changes associated with aging of the skin are manifested in xerosis, dramatic loss of skin elasticity due to damage to collagen and elastin fibers; as well as barrier function, modification of rhytides and deficiencies in the regenerative property of the skin. All of which ultimately result in thinning of the skin, malar fat atrophy and pigmentary changes. Autologous fat grafting or lipo injection containing stromal vascular fraction (SVF) acts like ideal soft tissue filler for facial filling and rejuvenation. It leads to progressive improvement of the skin texture, elasticity, and color over a few months, therefore adipose tissue seems to be not only a simple filler but also a dynamic filler with two types of different and supplementary effects, the volumetric effect and the regenerative effect.Cell assisted lipotransfer (CAL) is a technique that combines aspirated fat with concentrated ADSCs in the stromal vascular fraction (SVF) of the lipoaspirate. This technique could enhance the survival rate of the transplanted fat and leads to better cosmetic improvement

ELIGIBILITY:
Inclusion Criteria

1. Clinically diagnosed facial skin aging.
2. Glogau photoaging score II and III.
3. Body mass index ≥20 with adequate abdominal or other subcutaneous adipose tissue accessible for lipoaspiration.

Exclusion Criteria:

1. History of keloid formation.
2. Any coincidental chronic illness (e.g. metabolic, autoimmune or endocrinal) or malignancy.
3. Any bleeding or coagulation disorder or recent use of anticoagulant therapy.
4. Active infection.
5. History of any previous aesthetic procedure on the face within the past 6 months.
6. History of intake of anti-aging systemic or topical medications within the previous 3 months

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Assessment using hollowness severity rating scale :0 : no visible hollowness, 1: mild Hollowness, 2 : moderate Hollowness, 3: severe Hollowness | 3 months, 6 months
  serial photography for assessment using hollowness severity rating scale :0 : no visible hollowness, 1: mild Hollowness, 2 : moderate Hollowness, 3: severe Hollowness

SECONDARY OUTCOMES:
Measurement of hypodermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head | 3 months, 6 months
  Measurement of hypodermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head
Measurement of dermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head Measurement of dermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head | 3 months, 6 months
  Measurement of dermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Ibrahim Farid Mohammed Amin, MD, Study Director — Assistant Professor of Dermatology, Faculty of Medicine, Alexandria University.; Ossama Hussein Roshdy, MD, Study Director — Professor of Dermatology, Faculty of Medicine, University of Alexandria.; Wafaa Ibrahim Abdullah, MD, Study Director — Professor of Dermatology, Faculty of Medicine, University of Alexandria.; Radwa Ali Mehanna, PhD, Study Director — Assistant Professor of Physiology, Faculty of Medicine, Alexandria University; Nader Hussein Lotfy Bayoumi., MD, FRCS, Study Director — Professor of ophthalmology , Faculty of Medicine, University of Alexandria.
Locations (1):
- Aliaa Ismail, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roshdy OH, Abdallah WI, Farid CI, Mehanna RA, Bayoumi NH, Ismail AI. Stromal vascular fraction improves the durability of autologous fat temple augmentation-A split-face randomized study using ultrasound biomicroscopy. J Plast Reconstr Aesthet Surg. 2022 Jun;75(6):1870-1877. doi: 10.1016/j.bjps.2021.12.005. Epub 2022 Jan 15. PMID 35125305

DOCUMENTS (1):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03965936/Prot_000.pdf